CLINICAL TRIAL: NCT03282344
Title: A Pilot Study of NKTR-214 and Nivolumab in Selected Patients With Locally Advanced/Metastatic Sarcoma (CA209-9EM)
Brief Title: A Study of NKTR-214 in Combination With Nivolumab in Patients With Metastatic and/or Locally Advanced Sarcoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: M.D. Anderson Cancer Center (Other); Stanford University (Other); Rockefeller University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-366
Record Dates: First submitted 2017-09-12; First posted 2017-09-13 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: SARCOMA
Keywords: NKTR-214; NIVOLUMAB; 17-366
MeSH Terms: conditions — Sarcoma | interventions — bempegaldesleukin; Nivolumab

STUDY DESIGN:
Intervention Model Description: This is an open-label, multi-center, pilot study to evaluate the efficacy of NKTR- 214 in combination with nivolumab in patients with selected locally advanced/metastatic, high grade sarcoma.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- participants ≥18 years old NKTR-214 and Nivolumab (Experimental): NKTR-214 0.006mg/kg and nivolumab 360mg will be administered intravenously on day 1 of week 1 of cycle one and every 3 weeks (±3 days) thereafter.
  Interventions: Drug: NKTR-214; Drug: Nivolumab
- participants 12 - 17 years old NKTR-214 0.006mg/kg and Nivo (Experimental): NKTR-214 0.006mg/kg and nivolumab 360mg will be administered intravenously on day 1 of week 1 of cycle one and every 3 weeks (±3 days) thereafter.
  Interventions: Drug: NKTR-214; Drug: Nivolumab

INTERVENTIONS:
Drug: NKTR-214 — 0.006mg/kg IV on day 1 and every 3 weeks thereafter will be an intravenous (IV) infusion administered over 30 (±5) minutes every 3 weeks.
Drug: Nivolumab — 360mg (flat dose) IV infusion administered over 30 (±5) minutes every 3 weeks.

SUMMARY:
The purpose of this study is to test any good and bad effects of the combination of study drugs called NKTR-214 and nivolumab.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age ≥ 12 years at the time of informed consent
* Be capable, willing, and able to provide written informed consent/assent. For patients < 18 years of age, their parents or legal guardians must sign a written informed consent. Assent, when appropriate, will be obtained according to institutional guidelines.
* Be willing to comply with clinical trial instructions and requirements.
* Patients ≥ 18 years must be willing to comply with the mandatory biopsies.
* Patients must have a histologically confirmed metastatic and/or locally advanced sarcoma by the enrolling institution.
* For histological specific cohorts, patients must have confirmed metastatic and/or locally advanced osteosarcoma, chondrosarcoma, undifferentiated pleomorphic sarcoma/malignant fibrous histiocytoma high grade myxofibrosarcoma (UPS/MFH/MFS), vascular sarcoma, alveolar soft part sarcoma (ASPS), dedifferentiated/pleomorphic liposarcoma, Small Blue Round CellSynovial, or leiomyosarcoma (LMS) by the enrolling institution.

Note: Patients with confirmed sarcoma with histologies not defined by the above cohorts will be enrolled into the "Other" cohort.

* Adequate performance status:

  * Participants ≥16 years ECOG 0 or 1/KPS 100-70%
  * Participants <12-15 years Lanksky 100-70%
* Patients must have at least one prior line of systemic therapy (e.g.chemotherapy, immunotherapy, targeted or biological therapy) for their sarcoma if standard treatment is appropriate. Treatment naïve patients may be enrolled if they have refused standard systemic treatment. Prior adjuvant therapy will not count provided it was completed more than 6 months previously.
* Presence of measureable disease per RECIST v1.1.Target lesions must not be chosen from a previously irradiated field unless there has been radiographically and/or pathologically documented tumor progression in that lesion prior to enrollment.
* On echocardiogram, documented left ventricular ejection fraction >45%. Patients may instead have a multigated acquisition (MUGA) scan instead of transthoracic echocardiogram (TTE).
* Adequate organ function
* Women of childbearing potential (WOCBP) † must have a negative urine or serum pregnancy test at screening and ≤ 72 hours prior to day 1 of study treatment. If the urine pregnancy test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.

  † A woman of childbearing potential is a sexually mature female who: has not undergone a hysterectomy or bilateral oophorectomy; or has not been naturally postmenopausal for at least 24 consecutive months (i.e. has had menses at any time in the preceding 24 consecutive months).
* Male patients with WOCBP partners and female patients of childbearing potential must be willing to use an adequate method of contraception as outlined in Section 11.9, for the course of the study through 7 months (male participants) or 5 months (female participants) after the last dose of study medication.

Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the patient.

* Hematological

  * Absolute neutrophil count (ANC) ≥1,500 /mcL
  * Platelets ≥100,000 / mcL
  * Hemoglobin ≥9 g/dL or ≥5.6 mmol/L
* Renal

  * Serum creatinine OR Measured or calculateda creatinine clearance ≤1.5 X upper limit of normal (ULN) OR ≥60 mL/min for patient with creatinine levels > 1.5 X institutional ULN (GFR can also be used in place of creatinine or CrCl) Hepatic
  * Serum total bilirubin ≤ 1.5 X ULN OR Direct bilirubin ≤ ULN for patients with total bilirubin levels > 1.5 ULN
  * AST (SGOT) and ALT (SGPT) ≤ 2.5 X ULN OR ≤ 5 X ULN for patients with liver metastases
  * Albumin ≥ 2.5 mg/dL Coagulation
  * International Normalized Ratio [34] or Prothrombin Time [35]≤1.5 X ULN unless patient is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
  * Activated Partial Thromboplastin Time (aPTT) ≤1.5 X ULN unless patient is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants aCreatinine clearance should be calculated per institutional standard.

Exclusion Criteria:

* History of unstable or deteriorating cardiac disease within the previous 6 months prior to screening including but not limited to the following:

  * Unstable angina or myocardial infarction.
  * Congestive heart failure (New York Heart Association [NYHA] Class III or IV).
  * Uncontrolled clinically significant arrhythmias.
* Evidence of clinically significant interstitial lung disease or has known history of, or any evidence of active, non-infectious pneumonitis. .
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Patients with previously treated brain metastases may participate provided:

  * No current brain metastasis lesion greated than 2 cm. Patients with prior metastasis lesions greater than 2 cm that have been removed by surgical and/or radiotherapy may be enrolled if the lesion has been stable since surgery or radiotherapy.
  * No new or progressing brain metastatis of any size
  * No stereotactic radiation or craniotomy within 4 weeks of Cycle 1 Day 1
  * They are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment
  * No clinically signifigant symptoms secondary to brain metastases(This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.)
* Evidence of clinically significant immunosuppression such as the following:

  * Primary immunodeficiency state such as Severe Combined Immunodeficiency Disease
  * Concurrent opportunistic infection
  * Receiving systemic immunosuppressive therapy (> 2 weeks) including oral steroid doses > 10 mg/day of prednisone or equivalent within 2 months prior to enrollment. (Steroids for pre-medication for imaging studies are allowed.)
* History or evidence of symptomatic autoimmune disease (e.g., pneumonitis, glomerulonephritis, vasculitis, or other), or history of active autoimmune disease that has required systemic treatment (i.e., use of corticosteroids, immunosuppressive drugs or biological agents used for treatment of autoimmune diseases) in past 2 years prior to enrollment. Replacement therapy (e.g., thyroxine for hypothyroidism, insulin for diabetes or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment for autoimmune disease.
* Known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies) disease
* Patients known to be positive for active Hepatitis B (HBsAg reactive), or Hepatitis C (HCV RNA (qualitative) is detected)
* Prolonged QTcF > 450 ms for men and > 470 ms for women at Screening.
* Patients who have received a live vaccine within 30 days of the start date of the planned study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.
* Has a known history of active TB (Bacillus Tuberculosis)
* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
* Has a known history of active TB (Bacillus Tuberculosis)
* Is currently participating and receiving study therapy or using an investigational device or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 3 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

  * Note: Patients with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
  * Note: If patient received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapies.
* Hypersensitivity to nivolumab or any of its excipients.
* Hypersensitivity to NKTR-214 or any of its excipients.
* Need for > 2 antihypertensive medications for management of hypertension (including diuretics).
* Women who are pregnant or breast feeding

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2017-09-12 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
number of patients with a response | 2 years
  Primary Response Criteria (RECIST 1.1) Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progressions). Stable Disease [1]: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters whi le on study.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra D'Angelo, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Memorial Sloan Kettering Cancer Center (only recruiting to the Vascular/Angiosarcoma cohort), New York, New York
  - MD Anderson Cancer Center (only recruiting to the Vascular/Angiosarcoma cohort), Houston, Texas

REFERENCES:
- [Derived] D'Angelo SP, Richards AL, Conley AP, Woo HJ, Dickson MA, Gounder M, Kelly C, Keohan ML, Movva S, Thornton K, Rosenbaum E, Chi P, Nacev B, Chan JE, Slotkin EK, Kiesler H, Adamson T, Ling L, Rao P, Patel S, Livingston JA, Singer S, Agaram NP, Antonescu CR, Koff A, Erinjeri JP, Hwang S, Qin LX, Donoghue MTA, Tap WD. Pilot study of bempegaldesleukin in combination with nivolumab in patients with metastatic sarcoma. Nat Commun. 2022 Jun 16;13(1):3477. doi: 10.1038/s41467-022-30874-8. PMID 35710741
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm